CLINICAL TRIAL: NCT03228004
Title: Type 1 Diabetes Data Acquisition and Transfer Adherence Study
Acronym: T1D-DATA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201700818
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will be provided with training on how to upload glucose data via GLOOKO and will receive reminders to upload glucose data on a biweekly basis between clinic visits.
  Interventions: Behavioral: Glooko MeterSync

INTERVENTIONS:
Behavioral: Glooko MeterSync — The participant and caregiver will receive a reminder via text or email to upload glucose data via Glooko on a biweekly basis.

SUMMARY:
The purpose of this pilot study is to determine if training and support, combined with reminders to facilitate glucose data sharing with the diabetes care team in between clinic visits, can improve glycemic outcomes for patients ages 10-17 with type 1 diabetes who have HbA1c levels above target.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with T1D at least 6 months before consent is obtained
* Aged ≥ 2 years and ≤17 years at time of enrollment
* Must have access to a smartphone, tablet or computer at home with wireless connectivity
* Last HbA1c of ≥7.6% and ≤11%
* Using fixed doses, multiple daily injections or an insulin pump as primary diabetes management regimen
* Ability to read and speak English
* Patient at UF Health Pediatric Diabetes Clinic

Exclusion Criteria:

* Significant medical comorbidity in the child or adolescent that could, in the opinion of the PI, affect participant's capacity to complete study follow up
* Inability to read and speak English
* Not using insulin therapy
* Lack of access to mobile device or computer with wireless internet connectivity
* Unwilling or unable to use clinic's software (Glooko) to facilitate glucose data upload

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Improved glycemic control | 16 weeks
  HbA1c
Frequency of data upload | 16 weeks
  The number of times glucose data is uploaded between clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Albanese-O'Neill, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States